CLINICAL TRIAL: NCT06944249
Title: The Role of YAP1 in Fibrosis Explored Through Its Local Inhibition With Verteporfin in Surgical Wounds: A Randomized Controlled, Prospective, Evaluator-blinded Proof-of-concept Study.
Brief Title: Effect of YAP1-inhibition in Surgical Wounds.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jöri Pünchera (Other)
Collaborators: University of Geneva, Switzerland (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Jöri Pünchera, attending physician, M.D., University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CCER_Etude 2024- 00419
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Scar Formation
Keywords: YAP1; Verteporfin; Scar; Fibrosis; Wound healing
MeSH Terms: conditions — Cicatrix; Fibrosis | interventions — Verteporfin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study arm (verteporfin) (Experimental)
  Interventions: Drug: Verteporfin Injection
- Placebo arm (Placebo Comparator)
  Interventions: Drug: NaCl (placebo)

INTERVENTIONS:
Drug: NaCl (placebo) — During the safety margin excision, the placebo (NaCl) will be injected into the wound before suturing.
  Arms: Placebo arm
Drug: Verteporfin Injection — During the safety margin excision, the study drug (Verteporfin) will be injected into the wound before suturing.
  Arms: Study arm (verteporfin)

SUMMARY:
When we get injured, our body naturally tries to heal. In adults, this healing often leads to scars - thick, stiff tissue known as fibrotic tissue. Unlike normal tissue, fibrotic tissue doesn't function properly and can cause serious health problems, depending on the affected organ. Once it forms, fibrosis is usually permanent.

A good example of the fibrosis process is the healing of our skin: after a cut or surgery, the resulting scar is a type of fibrosis. Special cells called fibroblasts are key players in this process.

Our study looks at a drug called verteporfin, which is already approved both in Europe and the U.S. Previous research on mice and human cells suggests it can reduce or even prevent fibrosis.

We are now testing, clinically, histologically and by scRNA-seq, whether injecting verteporfin into the skin during wound healing, specifically after surgical procedures, can prevent thick, rigid scars from forming. Since the skin is easy to observe and sample, it offers a great model for studying this.

Will verteporfin have an impact on how surgical wounds heal? That's what we aim to find out.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent as documented by signature
* Age is >/= 18 years and < 56 years (differently said: starting from the 18th birthday to completion of their 55 years)
* Indication for a safety margin excision (5 mm laterally) due to melanoma in situ or severe dysplastic nevi previously completely excised
* Length of initial scar from 15 mm to 50 mm
* The initial lesion was excised on the back (to ensure that all patients undergo their safety margin excision within the internationally accepted timeframe, we will also accept patients requiring the procedure at another anatomical site if a particular batch cannot be filled within 4 weeks of its first patient's enrollment)

Exclusion Criteria:

* Clinical adenopathy (cervical, axillar, inguinal) defined as a lymph node of more than 1 cm diameter
* Melanoma in situ of lentigo maligna or acral lentiginous type
* Head and neck location
* Diameter of initial lesion above or equal to 3 cm
* Known and documented hypersensitivity to Verteporfin or to any of its excipients: lactose monohydrate, egg phosphatidylglycerol (to simplify we will exclude patients with known and documented allergy to egg protein), dimyristoyl phosphatidylcholine, ascorbyl palmitate, butylated hydroxytoluene (E321)
* Porphyria
* Moderate hepatic dysfunction referred to as any of the following: AST >1.2x upper normal range, ALT >1.2x upper normal range, decreased albumin level, prolongation of PT
* Biliary obstruction referred to as any of the following: ALP >1.2x upper normal range, GGT >1.2x upper normal range, anormal bilirubin level
* Pregnancy referred to as: positive beta-hCG blood test
* Breast-feeding
* Planned pregnancy in the next 6 months
* History of either one of the following: keloids, scleroderma, morphea, lupus erythematosus, nephrogenic systemic fibrosis, graft-versus-host disease, lichen sclerosus, eosinophilic fasciitis, Ehlers-Danlos syndrome, cutis laxa, Marfan syndrome, or pseudoxanthoma elasticum

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of the profibrotic mesenchymal fibroblast subpopulation in the study group compared to the placebo group. | There are 90 +/- 10 days between visit 1 and visit 4.
  For comparison between groups, skin samples of the repaired tissue taken at visit 4 (Day 90 +/- 10) will be compared between the patients of both groups.

SECONDARY OUTCOMES:
The changes of fibroblast subpopulations, clusters, and their different cell-cell interactions in both groups before and after the study intervention. | There are 90 +/- 10 days between visit 1 and visit 4.
  For comparison over time in both groups, skin samples of the repaired tissue taken at visit 4 (Day 90 +/- 10) will be compared to the scar sample of visit 1 (Day 0) in all patients of both groups.
Quantification of pilosebaceous units and profibrotic activity (quantity of collagen I and III and its ratio, fibronectin, α-SMA, nuclear localization of YAP1 and En1-staining) and its change over time | There are 90 +/- 10 days between visit 1 and visit 4.
  For comparison over time in both groups, skin samples of the repaired tissue taken at visit 4 (Day 90 +/- 10) will be compared to the scar sample of visit 1 (Day 0) in all patients of both groups.
Quantification of the different fibroblast subpopulations in unwounded, healthy skin. | The initial excision will take place 21 to 54 days before V1.
  In all patients, 2 slices of the initial FFPE skin samples will be analyzed.
The changes of different fibroblast subpopulations passing from unwounded skin to scarred, to repaired skin. | There are a maximum of 56 days + 90 +/- 10 days between the inital mole removal and visit 4.
  Analysis of the initial FFPE skin samples compared to the analysis on Day 0 and Day 90 (+/- 10).
Comparison of the clinical outcomes of the scars in both groups. | There are a minimum of 154 and a maximum of 178 days between visit 3 and visit 5.
  The clinical outcomes will be evaluated by VSS scoring at visit 3 (Day 14 +/- 2), visit 4 (Day 90 +/- 10) and visit 5 (Day 180 +/- 10).
The comparison of PROMs | There are a minimum of 154 and a maximum of 178 days between visit 3 and visit 5.
  PROMs will be assessed in both groups by SCAR-Q scoring at Day 14 (+/- 2), Day 90 (+/- 10) and Day 180 (+/- 10).

CONTACTS AND LOCATIONS:
Overall Officials: Jöri Pünchera, M.D., Principal Investigator — University Hospital, Geneva

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the assessment of primary and secondary outcomes, will be shared in a coded, anonymized format via a secure repository in accordance with FAIR data principles and Open Research Data guidelines. Data will be made available to qualified researchers upon reasonable request following publication. Access may be subject to a data use agreement.

REFERENCES:
- [Background] Mascharak S, desJardins-Park HE, Davitt MF, Griffin M, Borrelli MR, Moore AL, Chen K, Duoto B, Chinta M, Foster DS, Shen AH, Januszyk M, Kwon SH, Wernig G, Wan DC, Lorenz HP, Gurtner GC, Longaker MT. Preventing Engrailed-1 activation in fibroblasts yields wound regeneration without scarring. Science. 2021 Apr 23;372(6540):eaba2374. doi: 10.1126/science.aba2374. PMID 33888614
- [Background] Jiang D, Correa-Gallegos D, Christ S, Stefanska A, Liu J, Ramesh P, Rajendran V, De Santis MM, Wagner DE, Rinkevich Y. Two succeeding fibroblastic lineages drive dermal development and the transition from regeneration to scarring. Nat Cell Biol. 2018 Apr;20(4):422-431. doi: 10.1038/s41556-018-0073-8. Epub 2018 Mar 28. PMID 29593327
- [Background] Jiang D, Rinkevich Y. Converting fibroblastic fates leads to wound healing without scar. Signal Transduct Target Ther. 2021 Sep 1;6(1):332. doi: 10.1038/s41392-021-00738-6. No abstract available. PMID 34471094